CLINICAL TRIAL: NCT01166074
Title: Retrospective Chart Review Study: Subcutaneous IgG in Children Under 2 Years of Age
Brief Title: Retrospective Chart Review of Subcutaneous IgG Use in Infants
Status: Completed | Type: Observational
Sponsor: CSL Behring (Industry)
Responsible Party: Global Head Clinical Research & Development, CSL Behring
Other Study IDs: Ig_6001_R_D
Record Dates: First submitted 2010-07-19; First posted 2010-07-20 (Estimated); Last update posted 2011-02-11 (Estimated); Status verified 2011-02

CONDITIONS: Primary Immune Deficiency
MeSH Terms: conditions — Primary Immunodeficiency Diseases | interventions — Vivaglobin

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- SCIG
  Interventions: Biological: Subcutaneous IgG (SCIG)

INTERVENTIONS:
Biological: Subcutaneous IgG (SCIG) — Administered according to normal clinical practice
  Other Names: Vivaglobin; SCIG

SUMMARY:
This study is a retrospective chart review of the use of subcutaneous IgG (SCIG) in infants less than two years old.

ELIGIBILITY:
Inclusion Criteria:

* Infants who received more than one dose of IgG by the subcutaneous route before the age of two years.
* Consent of parent/guardian if required by institution/IRB.

Exclusion Criteria:

* Infants with protein losing conditions such as lymphangiectasis, nephrosis, S/P cardio-thoracic surgery requiring drainage tubes for more than 48 hrs, protein losing enteropathy.
* Concomitant treatment with plasma, other blood products or IGIV while on SCIG.
* Lack of consent by parent/guardian (if required by Institution/IRB).
* Any other condition or treatment which, in the opinion of the local investigator, would interfere with obtaining valid results for that subject.

Max Age: 2 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: Children under 2 years of age
Sampling Method: Non-Probability Sample
Enrollment: 27 (Actual)
Dates: Start 2010-05; Primary Completion 2010-12 (Actual); Study Completion 2010-12 (Actual)

PRIMARY OUTCOMES:
SCIG use | 1 year
  To describe the use of SCIG in infants below the age of two years in major academic medical centers and immunologists' practices in the US

SECONDARY OUTCOMES:
Number of infants who received more than one dose of SCIG, then continued receiving IgG by a route other than SC | 1 year

CONTACTS AND LOCATIONS:
Overall Officials: Melvin Berger, MD, PhD, Principal Investigator — CSL Behring
Locations (5):
- United States (5):
  - Children's Hospital of Los Angeles, Los Angeles, California
  - University of South Florida, Tampa, Florida
  - Midwest Immunology Clinic, Plymouth, Minnesota
  - University Hospitals Case Medical Center, Cleveland, Ohio
  - St. Judes Children's Research Hospital, Memphis, Tennessee